CLINICAL TRIAL: NCT00420433
Title: Prospective Study of Tumor Response Assessment in Metastatic Breast Cancer Involving Bones
Brief Title: Bone Response in Metastatic Breast Cancer Involving Bones
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-0999
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer; Bone Metastases
Keywords: Breast Cancer; Bone Metastases; Radiography; X-Ray; Computed Tomography; CT Scan; Skeletal Scintigraphy
MeSH Terms: conditions — Breast Neoplasms | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with breast cancer that has spread to the bones.
  Interventions: Procedure: Skeletal Scintigraphy; Procedure: Radiography; Procedure: CT Scan

INTERVENTIONS:
Procedure: Skeletal Scintigraphy — Performed before treatment and again at 3, 6, 9, and 12 months after starting anticancer therapy.
Procedure: Radiography — Performed before treatment and again at 3, 6, 9, and 12 months after starting anticancer therapy.
  Other Names: X-Ray
Procedure: CT Scan — CT scan will include your chest, abdomen, and pelvis. Performed before treatment and again at 3, 6, 9, and 12 months after starting anticancer therapy.
  Other Names: Computed Tomography

SUMMARY:
Primary Objectives:

* To estimate and compare the sensitivity and specificity of computed tomography (CT), plain radiography (XR), and skeletal scintigraphy (SS) with each other for the assessment of response of bone metastasis in patients with breast cancer.
* To estimate and compare the sensitivity and specificity of M. D. Anderson (MDACC) bone metastasis criteria with that of current criteria (UICC, WHO) in breast cancer patients for the assessment of the behavior of osseous metastasis in breast cancer patients.

Secondary Objective:

* To evaluate the progression free survival (PFS) and overall survival (OS) of each response group (CR, PR, SD, PD) assessed by imaging and response criteria.

DETAILED DESCRIPTION:
This study will compare plain x-rays (XR), skeletal scintigraphy (SS), computed tomography (CT), magnetic resonance imaging (MRI), and positron emission tomography/CT (PET/CT) in measuring response. MRI and PET/CT can be performed if they are needed by standard of care. We anticipate MRI will be performed most commonly due to back pain.

Researchers will also compare three sets of standardized evaluation criteria (UICC criteria, WHO criteria, MDACC criteria). The MDACC criteria are new while the UICC and the WHO are standard criteria. The old criteria are no longer thought to be as reliable because they are based only on older technology (XR and SS). Since newer technologies are not included in the old criteria, most cancer doctors do not use these older criteria for evaluation of bone lesions. Therefore, new bone tumor criteria including newer imaging techniques (CT and MRI) are needed. At the end of the study, researchers will look at how sensitive and clear each imaging technique is, and they will use a set of criteria to learn which technique best measures the disease's response to therapy.

Participants in this study will have a complete physical exam, including a score of their bone pain. Routine blood tests (between 1-2 tablespoons) will be performed before participation in this study begins. Women who are able to have children must have a negative blood pregnancy test before starting treatment.

Participants will also have imaging examinations (XR, SS, CT, and MRI, PET/CT).

All of the first examinations will be finished within one month before the start the anti-cancer therapy. If imaging examinations alone cannot prove that the disease has spread to the bone, a needle bone biopsy will be done. A bone biopsy means that researchers will collect a couple of small tumor samples from the suspicious bone site. The tumor samples will be taken using a large needle while you are under the appropriate anesthesia.

If you are found to be eligible for this study, you will have imaging exams (described below), bone score evaluations, and blood tests (between 1-2 tablespoons) done before treatment and again at 3, 6, 9, and 12 months after starting anticancer therapy.

Plain radiographs:

Also called X-rays. You will receive a complete bone survey. This consists of 2 views of spine, one view of the top of your head, one view of your chest, one view of your pelvic bones, and two of your ribs, one from each side. Any other symptomatic bone scans will also be included.

Skeletal scintigraphy:

Also called bone scan. You should not eat for more than 4 hours before this examination. You will get the pictures 2-3 hour after intravenous injection of Technetium-99m bound to methylene diphosphonate (Tc-99m MDP).

CT:

CT scan will include your chest, abdomen, and pelvis. You should not eat for more than 6 hours before this examination. You will be given oral and intravenous contrast as is done in standard care.

MRI:

This is an optional procedure. MRI of the symptomatic areas will be performed and followed on the same schedule as other imaging. You will be given contrast dye by vein as is done in standard care.

PET/CT:

This is an optional procedure. The examination usually takes 30-40 min while you are lying on the moving bed with tunnel 60-90min after injection of 2-deoxy-2-[18F] fluoro-D-glucose (FDG) by vein. You should not eat for more than 6 hours before this examination.

Your part in the study will end after the 12 month tests. However, you will be monitored for 3 years after enrolling on this study.

This is an investigational study. This study is not focusing to test the treatment agents but to test the imaging technique assessing bone tumor response. The exams performed in this study are commercially available and are part of routine examination. A total of up to 120 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed bone (from calvarium to pelvis include ribs and sternum) and nonosseous (it should be measurable by CT) metastasis or primary breast tumor (with a confirmation of no surgical treatment for 12 months) from breast cancer. If the bone metastasis is not confirmed by imaging, bone biopsy is needed. Please see diagnostic flow sheet. (APPENDIX B)
2. Zubrod performance status 2 or less. (APPENDIX A)
3. Patient must receive systemic treatment (e.g., chemotherapy, hormonal therapy) for this newly diagnosed metastatic disease. (Additional bisphosphonate treatment will be acceptable.)
4. Patients must sign an informed consent document indicating awareness that this study is not focusing on the verification of treatment agents but on verification of modalities to assess bone tumor response, in keeping with institutional policy.

Exclusion Criteria:

1. Patients who have less than 3 months interval from completion of treatment (chemotherapy and/or radiation therapy) for primary breast cancer.
2. Patients who have the history of radiation therapy for bone disease.
3. History or presence of brain/leptomeningeal metastasis.
4. History of other malignancies except cured non-melanoma skin cancer or cured cervical carcinoma in situ

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants with breast cancer that has spread to the bones.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To compare different imaging techniques in measuring the response of bone disease to treatment. | 5 Years

SECONDARY OUTCOMES:
To compare different evaluation techniques (evaluation criteria) in reading the images. | 5 Years
To study the change in the response of blood serum markers and the reliability of biochemical markers. | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org